CLINICAL TRIAL: NCT05842447
Title: Effect of Two Doses of Pomanox® Pomegranate Extract Consumption on Skin Ageing. Randomized, Parallel, Placebo Controlled and Triple Blind Clinical Trial (POMASKIN).
Brief Title: Effect of Pomanox® on Skin Ageing (POMASKIN)
Acronym: POMASKIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: Euromed, S.A. (Unknown)
Responsible Party: Principal Investigator, Antoni Caimari, Director of Eurecat's Biotechnology Area, Fundació Eurecat
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: POMASKIN
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Skin Ageing
Keywords: Photoageing; Polyphenols; Natural extracts; Collagen metabolism; Hyaluronic acid; Oxidative stress; Antiglycan effect; Inflammatory system; Intestinal microbiota; skin microbiota
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 367 mg Pomanox group (Experimental): One capsule daily with 367 mg of Pomanox®P30 for 12 weeks
  Interventions: Dietary Supplement: 367 mg Pomanox group
- 700 mg Pomanox group (Experimental): One capsule daily with 700 mg of Pomanox®P30 for 12 weeks
  Interventions: Dietary Supplement: 700 mg Pomanox group
- Control group (Placebo Comparator): One capsule daily with maltodextrin for 12 weeks
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: 367 mg Pomanox group — Treatment with 367 mg Pomanox®P30 during 12 weeks
  Arms: 367 mg Pomanox group
Dietary Supplement: 700 mg Pomanox group — Treatment with 700 mg Pomanox®P30 during 12 weeks
  Arms: 700 mg Pomanox group
Dietary Supplement: Control group — Treatment with maltodextrin during 12 weeks
  Arms: Control group

SUMMARY:
The state of skin health impacts not only on the general health of individuals, but also on mental health. Ultraviolet radiation (UV) is one of the main external factors that causes skin ageing, producing photo-aging, characterized by multiple alterations in the skin such as the appearance of wrinkles, dryness, erythema, alterations in the pigmentation, inflammation and increased fragility.

Several studies show that polyphenols extracts, including pomegranate extracts, have beneficial effects on various skin characteristics induced by photoaging by modulating internal factors that lead to changes associated with photoaging. Among these internal factors are oxidative stress, glycation stress caused by an accumulation of advances glycation end-products (AGEs), inflammation, and the composition of the intestinal and skin microbiota.

Pomanox® is a polyphenolic extract derived from pomegranate for which antioxidant activity and positive effects on the metabolism of collagen and hyaluronic acid have been shown in previous in vitro studies.

DETAILED DESCRIPTION:
The hypothesis of the study is that the consumption of Pomanox®P30 will have beneficial effects on skin ageing in humans through the modulation of the metabolism of collagen, hyaluronic acid and the inflammatory system, the inhibition of the production of reactive oxygen species and AGEs, and/or changes in the intestinal and skin microbiota composition.

The main objective of the study is to evaluate the effect of consuming two doses of Pomanox®P30 on hyperpigmented skin spots in humans.

The secondary objectives of the study are to evaluate the effects of consuming two doses of Pomanox®P30 on other parameters related to skin ageing (wrinkles, elasticity, erythema index, hydration, pores, acne and keratin), on different markers of collagen and hyaluronic acid metabolism, oxidative stress, the anti-glycan effect and the inflammatory system, and on the composition of the intestinal and skin microbiota.

A randomized, parallel, placebo-controlled, single-center, triple-blind clinical trial with a 1:1:1 ratio between interventions with 66 participants will be conducted.

Each participant will make 4 visits:

* A pre-selection visit (to check inclusion/exclusion criteria) (V0), and if the eligibility criteria are met,
* 3 study visits during the consumption of the treatments, which will take place on the first day of the study (V1), at 29 days of treatment (V2) and at 85 days of treatment (V3).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30 years or older and 65 years or less.
* Fitzpatrick skin phototype II-IV.
* Read, write and speak Catalan or Spanish.
* Sign the informed consent.

Exclusion Criteria:

* Present any chronic gastrointestinal disease that may interfere with the objectives of the study such as celiac disease, Crohn's disease, ulcerative colitis, irritable bowel syndrome with symptoms in the last 6 months, chronic diarrhea, or having undergone any bariatric surgery procedure.
* Present a chronic disease with clinical manifestation and/or being under pharmacological treatment that may interfere with participation in the study.
* Present values of body mass index ≥ 35 kg/m^2.
* Present a clinical history of active anemia.
* Have consumed or intended to consume during the study treatments, supplements or multivitamin supplements or phytotherapeutic products that interfere with the study treatment (such as retinol or vitamin A, vitamin C, vitamin E, antioxidants, polyphenols, probiotics and prebiotics) up to 30 days before the start of the study intervention.
* Have consumed or intended to consume during the study contraceptive treatments or hormonal therapy up to 30 days before the start of the study intervention.
* Have taken treatment with antibiotics up to 30 days before the start of the study intervention.
* Have taken or intended to take treatments for acne, for photo-ageing or to improve the appearance or condition of the skin (such as chemical peeling, laser therapy, light therapy or hyaluronic acid injection; regular treatment in a facial beauty salon, skin whitening agents) up to 6 months before the start of the study intervention.
* Being a smoker or ex-smoker in the last 6 months before inclusion in the study.
* Consume 2 o more Standard Beverage Units daily or 17 weekly.
* Present allergy and/or intolerance to the study products (such as presenting hypersensitivity to maltodextrin or allergy to pomegranate).
* Being pregnant or intending to become pregnant.
* Being in breastfeeding period.
* Being participating, intending to participate or having participated in a clinical trial or nutritional intervention study in the last 30 days before inclusion in the study.
* Present any skin disease (such as atopic skin, eczema, neurodermatitis, vitiligo or psoriasis) or any skin disorder in the sudy area (such as irritations, moles, scars or macules).
* Have been intensely exposed to the sun or artificial ultraviolet radiations (solarium) in the test area during the 30 days before the start of the study or planning to do so during the study.
* Not being able to follow the guidelines of the study.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Change in skin melanin index. | At day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Skin melanin index measured by using a Mexameter® MX18.

SECONDARY OUTCOMES:
Change in skin wrinkles. | At day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Skin wrinkles measured using a DermoPrime System.
Change in skin hydratation. | At day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Skin hydratation measured using a DermoPrime System.
Change in skin elasticity. | At day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Skin elasticity measured using a Cutometer ®MPA 580.
Change in skin erythema index. | At day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Skin erythema index measured by using a Mexameter® MX18.
Change in skin pores. | At day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Skin pores measured using a DermoPrime System.
Change in skin acne. | At day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Skin acne measured using a DermoPrime System.
Change in skin keratin. | At day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Skin keratin measured using a DermoPrime System.
Change in Human Procollagen I N-Terminal Propeptide blood levels. | At day 1 (visit V1) and day 85 (visit 3).
  Serum levels of Human Procollagen I N-Terminal Propeptide will be measured using human ELISA kits.
Change in Human Procollagen I C-Terminal Propeptide blood levels. | At day 1 (visit V1) and day 85 (visit 3).
  Serum levels of Human Procollagen I C-Terminal Propeptide will be measured using human ELISA kits.
Change in Metalloproteinase-1 blood levels. | At day 1 (visit V1) and day 85 (visit 3).
  Serum levels of Metalloproteinase will be measured using human ELISA kits.
Change in hyaluronic acid blood levels. | At day 1 (visit V1) and day 85 (visit 3).
  Serum levels of hyaluronic acid will be measured using human ELISA kits.
Change in superoxide dismutase activity blood levels. | At day 1 (visit V1) and day 85 (visit 3).
  Serum superoxide dismutase activity will be measured using a colorimetric kits.
Change in reduced gluthathione blood levels. | At day 1 (visit V1) and day 85 (visit 3).
  Serum levels of reduced gluthathione will be measured using human ELISA kits.
Change in pentosidine blood levels. | At day 1 (visit V1) and day 85 (visit 3).
  Serum levels of pentosidine will be measured using human ELISA kits.
Change in carboxymethyl-lysine blood levels. | At day 1 (visit V1) and day 85 (visit 3).
  Serum levels of carboxymethyl-lysine will be measured using human ELISA kits.
Change in interleukin-1 alpha blood levels. | At day 1 (visit V1) and day 85 (visit 3).
  Serum levels of interleukin-1 alpha will be measured using human ELISA kits.
Change in interleukin-6 blood levels. | At day 1 (visit V1) and day 85 (visit 3).
  Serum levels of interleukin-6 will be measured using human ELISA kits.
Change in stool microbiota composition. | At day 1 (visit V1) and day 85 (visit 3).
  Total DNA extracted from stool samples will be sequenced on an Ion Torrent platform. It will be analysed the taxonomic profile, alpha diversity and beta diversity.
Change in skin microbiota composition. | At day 1 (visit V1) and day 85 (visit 3).
  Total DNA extracted from stool samples will be sequenced on an Ion Torrent platform. It will be analysed the taxonomic profile, alpha diversity and beta diversity.
Change in dimethylellagic acid glucuronide urine levels. | At day 1 (visit V1) and day 85 (visit 3).
  Urine levels of dimethylellagic acid glucuronide will be measured by Liquid Chromatography Mass Spectrometry.
Change in urolithin A glucuronide urine levels. | At day 1 (visit V1) and day 85 (visit 3).
  Urine levels of urolithin A glucuronide will be measured by Liquid Chromatography Mass Spectrometry.
Subject self-assessment quality of the skin. | At day 29 (visit V2) and day 85 (visit 3).
  The quality of the skin of the volunteers will be evaluated subjectively through self-assessment questionnaire of the subjects themselves. This questionnaire will assess the perception of the volunteers on the improvement of their skin in general and on wrinkles, spots, redness, elasticity, hydration, pores and acne. In the questionnaire there will be 5 grades to asses the state: worsened (0), slightly worsened (1), no change (2), slightly improved (3) and improved (4).
Age. | At day -7 (pre-selection visit).
  The age of the volunteers will be recorded in the case report form.
Height. | At day -7 (pre-selection visit).
  Height measured by a standardized method.
Change in body weight. | At day -7 (pre-selection visit), day 1 (visit V1, day 29 (visit 2) and day 85 (visit 3).
  Body weight measured by a standardized method.
Change in body mass index. | At day -7 (pre-selection visit), day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Weight and height will be combined to report Body Mass Index in kg/m^2.
Change in fat mass. | At day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Fat mass measured by TANITA SC 330.
Change in muscle mass. | At day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Muscle mass measured by TANITA SC 330.
Concomitant medication. | At day -7 (pre-selection visit), day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Concomitant medication consumed during the study will be recorded in the case report form.
Dietary supplements consumed. | At day -7 (pre-selection visit), day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Dietary supplements consumed during the study will be recorded in the case report form.
Use of cosmetic treatments. | At day -7 (pre-selection visit), day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  The use of cosmetic treatments during the study will be recorded in the case report form.
Exposure to ultraviolet radiation. | At day -7 (pre-selection visit), day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Exposure of volunteers to ultraviolet radiation will be recorded in the case report form.
Products with pomegranate and ellagitannins consumption. | At day -7 (pre-selection visit), day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Consumption of products with pomegranate and ellagitannins during the study will be recorded in the case report form.
Eating habits. | At day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Eating habits of volunteers during the study will be recorded using a food frequency questionnaire.
Physical activity. | At day 1 (visit V1), day 29 (visit 2) and day 85 (visit 3).
  Physical activity of volunteers during the study will be recorded using the international physical activity questionnaire.
Intervention compliance. | At day 29 (visit 2) and day 85 (visit 3).
  The intervention compliance by the volunteers will be assessed by counting the number of remaining capsules and applying the formula (Number of capsules consumed/Number of capsules to consume)x100.
Adverse events. | At day 29 (visit 2) and day 85 (visit 3).
  Possible adverse events derived from taking study's products will be recorded in the case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Caimari, PhD, Principal Investigator — Fundació Eurecat
Locations (2):
- Spain (2):
  - Anna Crescenti, Reus, Catalonia. Spain
  - Eurecat, Reus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org